CLINICAL TRIAL: NCT03339037
Title: Application of Hyperbaric Oxygen Therapy for Children Suffering From Prolonged Post-Concussion Syndrome Due to Mild Traumatic Brain Injury
Brief Title: Hyperbaric Oxygen Therapy Effect on Post Concussion Syndrome in Children
Acronym: TBIPED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties - patients refusal to sham controlled
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0120-16-ASF
Record Dates: First submitted 2017-10-22; First posted 2017-11-13 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Hyperbaric Oxygen Therapy; Traumatic Brain Injury; Post-Concussion Syndrome
Keywords: HBOT; TBI; pediatrics; PCS; PPCS; concussion; traumatic brain injury; hyperbaric oxygen
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome; Brain Concussion | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: randomized controlled trial using a SHAM treatment compared to treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomization by computer, sham/ treatment will be known to chamber technicians and nurses but not to investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric oxygen therapy (Active Comparator): 60 Hyperbaric oxygen sessions in a multiplace hyperbaric chamber (HAUX-Life-Support GmbH). each session 1.5 ATA of 100% oxygen for 1 hour.
  1 meter per minute compression and decompression.
  Interventions: Device: Hyperbaric oxygen therapy
- Normobaric air SHAM (Sham Comparator): 60 sessions in a multiplace hyperbaric chamber (HAUX-Life-Support GmbH). Each session at 1 ATA of 21% oxygen (air) for 1 hour.
  1 meter per minute compression and decompression. after 3 months, patients will be crossed over and treated with 60 sessions of treatment
  Interventions: Device: Normobaric air SHAM

INTERVENTIONS:
Device: Hyperbaric oxygen therapy — 60 HBOT sessions at 2 ATA 100% oxygen
  Arms: Hyperbaric oxygen therapy
Device: Normobaric air SHAM — 60 sessions at 1 ATA 21% oxygen (air)
  Arms: Normobaric air SHAM

SUMMARY:
Due its high incidence, mTBI and its consequences of PPCS are a major public health issue. There is no consensus regarding the treatment of PPCS in pediatrics. Relying on its results in adults, HBOT offers a promising new direction of treatment, which targets the basic pathological processes responsible for post-concussion symptoms.

The effect of hyperbaric oxygen therapy in pediatric TBI has never been evaluated.

The aim of the current study is to evaluate in a prospective cross-over, randomized study, the effect of HBOT on children with PPCS due to mild TBI.

DETAILED DESCRIPTION:
The study is designed as a prospective, randomized, controlled, cross-over two groups trial. The study will be conducted in the -Sagol center for hyperbaric medicine and research and the children neurological unit of Assaf Harofeh Medical Center, Israel. Brain MRIs evaluation will be done the radiology department of Assaf-Harofeh Medical Center, Israel.

Study will include 70 patients After signing the informed consent (signed by the parents), patients will undergo computerized cognitive tests using the computerized Neurotrax and Moxo cognitive batteries. Patients who fulfill inclusion criteria will be included in the study.

After signing informed consent (by parents, at the prescreening phase), patients who fill inclusion criteria, will be randomized in 1:1 manner into the treated or the control-cross group. Randomization will be performed using a computer software according to patient id. After the randomization, patients will be invited for baseline evaluation that will include full review of their medical status and complete physical examination.

All patients will go through evaluation of their neurocognitive function using further neurocognitive testing battery, questionnaires and brain imaging (perfusion MRI+DTI, SPECT). In cases of brain tumors, skull base tumors, encephalomalacia findings in MRI, patients will be excluded.

The patients in the treated group will be evaluated three time - at baseline, after 3 months of HBOT treatment and after another consequent 3 months period from treatment (6 months from baseline). The patients of the cross group will be evaluated three times as well- at baseline, after 3 month control period without hyperbaric treatment and after a consequent 3 month period of HBOT treatment.

The following HBOT treatment protocol will be practiced: The patients will go through 60 HBOT treatments (each treatment session will be given on a separate day), distributed over three months (five days a week). Each session will be for 60 minutes in 100% oxygen atmosphere and at pressure of 1.5 ATA.

ELIGIBILITY:
Inclusion Criteria:

* - Ages 8-15
* Mild TBI (defined as loss of consciousness with duration of 0-30 minutes, post-traumatic amnesia with duration of less than 24 hours, Glasgow Coma Scale grade of 13-15) within 6 months-3 years prior to the inclusion in the study.
* Moderate TBI -Patients with a GCS of 9-12 a as well as additional criteria such as CT abnormalities and admission to hospital
* Presence of at least two PCS as measured by the Post-Concussion Symptom Inventory )see attached) (there's a RCT now recruitingwith at least 1 and not 2) for at least 3 months.
* No change in cognitive or behavioral functions during one month prior to the beginning of the study (according to parents/teachers report).

Screening protocol:

After signing the informed consent (signed by the parents), patients will undergo computerized cognitive tests using the computerized Neurotrax in patients over 10, and standard pen and paper cognitive tests in patients under 10. Patients who fulfill inclusion criteria will be included in the study.

Inclusion criteria:

- Objective cognitive impairment: a decrease of at least 1 standard deviation (SD) from same age mean score in one or more of the following indices : memory, attention, information processing speed, executive functions in both Neurotrax

Exclusion Criteria:

* - Dynamic neurologic improvement or worsening during the past month (according to parents/teachers report);
* Had been treated with HBOT for any other reason prior to their inclusion;
* Chest pathology incompatible with pressure changes (including asthma)
* Inner ear disease;
* Claustrophobia;
* Inability to perform awake brain MRI test
* Previous neurologic conditions (eg. Epilepsy, neuromuscular diseases, metabolic diseases, etc.)
* Brain tumors
* Skull base fractures
* Active malignancy
* s/p neurosurgery that included: ventricular drainage, subdural hematomas drainage, epidural hematomas drainage, intracerebral hemorrhage evacuation. Depressed fracture surgery, won't be excluded.
* Encephalomalacia per MRI imaging
* No informed consent

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Cognitive function | at 3 months
  General,Attention, Memory, Executive functions, Visual spatial and Verbal memory indices Index (scale 0-100) will be measured using the computerized standardized Neurotrax battery test. Each of above cognitive indices is computed as a normalized combined score of 2-3 cognitive tests. (At baseline, this battery will be conducted as part of the screening in patients over 10).
Cognitive function | at 6 months
  General,Attention, Memory, Executive functions, Visual spatial and Verbal memory indices Index (scale 0-100) will be measured using the computerized standardized Neurotrax battery test. Each of above cognitive indices is computed as a normalized combined score of 2-3 cognitive tests. (At baseline, this battery will be conducted as part of the screening in patients over 10).

SECONDARY OUTCOMES:
Post concussion syndrome symptoms | baseline, 3 months and 6 months from baseline
  Patients and their parents will fill questionaries' Postconcussion Symptom Inventory (PCSI) (scale 0-21) at baseline and at their second and/or third evaluations
Health Behaviour inventory | baseline, 3 months and 6 months from baseline
  Patients and their parents will fill questionaries' Health Behaviour inventory (scale 50-200) at baseline and at their second and/or third evaluations
Balance | baseline, 3 months and 6 months from baseline
  Patients will undergo balance tests (BERG Balance Scale) (scale 0-56) at each of the evaluations
Brain functional imaging | baseline, 3 months
  Patients will undergo photon emission tomography (PET-CT) using FDG at each of the three evaluations
Brain microstructural imaging | baseline, 3 months and 6 months from baseline
  Imaging will be conducted in using a 3 Tesla system (Siemens, Germany). The MRI protocol includes the following sequences: Axial T1, T2, FLAIR, Axial Diffusion weighted, Axial T1-PostGadollinium , dynamic contrast enhancement (DSC), diffusion tensor imaging (DTI)
Brain perfusion | baseline, 3 months and 6 months from baseline
  Imaging will be conducted in using a 3 Tesla system (Siemens, Germany). The MRI protocol includes the following sequences: Axial T1, T2, FLAIR, Axial Diffusion weighted, Axial T1-PostGadollinium , dynamic contrast enhancement (DSC), diffusion tensor imaging (DTI)
Short form health survey (PedsQL) | baseline, 3 months and 6 months from baseline
  Patients and their parents will complete questionnaires Pediatric Quality of Life inventory (PedsQL) - multi-dimensional concept that includes domains related to physical, mental, emotional, and social functioning.
Brain network analysis | baseline, 3 months and 6 months from baseline
  Patients will undergo resting state EEG as well as EEG during performing cognitive tasks ,using a 64 electrodes cap.
Behaviour | baseline, 3 months and 6 months from baseline
  The parents and their teachers will complete the following questionnaire at baseline and at their second and/or third evaluations. The rating scales are available for parent (Conners 3-P), teacher (Conners 3-T) and self-report (Conners 3-SR).Subscales include inattention, hyperactivity/impulsivity, learning, executive functioning, aggression and peer relations, as well as subscales mapping onto DSM-IV criteria for ADHD (inattentive), ADHD (hyperactive-impulsive), ADHD combined, Conduct Disorder, and Oppositional-Defiant Disorder. Means and standard deviations for the global index vary dependent on age (for 6 year-olds the mean is 5.15 with a standard deviation of 3.97; means for 17 to 18 year-olds are 3.90 with a standard deviation of 4.00). Raw scores are usually converted to T-scores or percentile scores relative to normative data. T-scores above 60 (percentiles above 84) are considered clinically significant.
Executive functions | baseline, 3 months and 6 months from baseline
  The parents and their teachers will complete the Behavior Rating Inventory of Executive Function(BRIEF) questionnaire at baseline and at their second and/or third evaluations.
  he Global Executive Composite (GEC) is an overarching summary score that incorporates all of the BRIEF clinical scales. The possible range of scores for teachers is 0 to 24.

CONTACTS AND LOCATIONS:
Overall Officials: Shai a Efrati, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No